CLINICAL TRIAL: NCT00910715
Title: Duration of Antibiotic Treatment of Erythema Migrans. A Randomized Clinical Trial.
Brief Title: Duration of Antibiotic Treatment of Erythema Migrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Franc Strle, M.D., PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EM-0509
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Erythema Chronicum Migrans
Keywords: erythema migrans; Lyme borreliosis; doxycycline treatment; outcome; subjective symptoms
MeSH Terms: conditions — Erythema Chronicum Migrans; Glossitis, Benign Migratory; Lyme Disease | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EM-10 days doxycycline (Active Comparator)
  Interventions: Drug: doxycycline
- EM-doxycycline 15 days (Active Comparator)
  Interventions: Drug: doxycycline
- controls (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: doxycycline — doxycycline 100 mg bid, 10 days
  Arms: EM-10 days doxycycline
Drug: doxycycline — doxycycline 100 mg bid, 15 days
  Arms: EM-doxycycline 15 days
Drug: placebo — control subjects without a history of Lyme borreliosis
  Arms: controls

SUMMARY:
The purpose of this study is to compare the efficacy of 15-day versus 10-day doxycycline treatment in patients with erythema migrans.

ELIGIBILITY:
Inclusion Criteria:

* solitary erythema migrans in patients > 15 years

Exclusion Criteria:

* a history of Lyme borreliosis in the past
* pregnancy or lactation
* immunocompromised status
* serious adverse event to doxycycline
* taking antibiotic with antiborrelial activity within 10 days
* multiple erythema migrans or extracutaneous manifestations of Lyme borreliosis

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD, Study Chair — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia

REFERENCES:
- [Derived] Veluscek M, Bajrovic FF, Strle F, Stupica D. Doxycycline-induced photosensitivity in patients treated for erythema migrans. BMC Infect Dis. 2018 Aug 3;18(1):365. doi: 10.1186/s12879-018-3270-y. PMID 30075748
- [Derived] Stupica D, Lusa L, Ruzic-Sabljic E, Cerar T, Strle F. Treatment of erythema migrans with doxycycline for 10 days versus 15 days. Clin Infect Dis. 2012 Aug;55(3):343-50. doi: 10.1093/cid/cis402. Epub 2012 Apr 20. PMID 22523260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients older than 15 years evaluated between June and October 2009 at the Lyme Borreliosis Outpatient Clinic, University Medical Center Ljubljana, Slovenia were eligible for the study if they had typical solitary erythema migrans as defined by CDC.
  Patients were asked to refer a spouse/friend of the same age ± 5 years to serve as a control.
Pre-assignment Details: 241 were evaluated for enrollment and not enrolled in the study.
Groups:
- EM-10 Days Doxycycline: doxycycline 100 mg b.i.d. for 10 days
- EM-doxycycline 15 Days: doxycycline 100 b.i.d. for 15 days
- Controls: subjects without a history of Lyme borreliosis included in the study at the 6 month follow-up time point
Period: Overall Study
Arm/Group | EM-10 Days Doxycycline | EM-doxycycline 15 Days | Controls
Started | 108 | 117 | 81
Completed | 86 | 91 | 81
Not Completed | 22 | 26 | 0
Not completed — Lost to Follow-up | 22 | 26 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EM-10 Days Doxycycline | EM-doxycycline 15 Days | Controls | Total
Number analyzed (Participants) | 108 | 117 | 0 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 |  | 4
  Between 18 and 65 years | 88 | 101 |  | 189
  >=65 years | 18 | 14 |  | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (14.3) | 49.6 (14.0) |  | 50.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 63 |  | 125
  Male | 46 | 54 |  | 100
Region of Enrollment [Number; unit: participants]
  Slovenia | 108 | 117 |  | 225

OUTCOME MEASURES:

1. Primary Outcome: Objective Sequelae and Post-treatment Subjective New or Increased Symptoms (NOIS)in Patients Treated for Erythema Migrans With Doxycycline for 10 or 15 Days.
Description: At each visit patients were examined and asked about the presence of any symptoms that newly developed/had worsened since erythema migrans. If such symptoms had no other medical explanation they were regarded as new or increased symptoms (NOIS). Complete response=absence of any manifestations of Lyme borreliosis, with return to pre-Lyme borreliosis health status. Partial response=presence of NOIS. Failure=presence of objective manifestations of Lyme borreliosis or persistence of B. burgdorferi sensu lato in skin at the site of the previous erythema migrans.
Time Frame: 1 year follow-up
Population: Number of participants with complete response to treatment.
Measure: Number; unit: number of participants
Groups:
- Controls: subjects without a history of Lyme borreliosis included in the study as controls only at the 6 month follow-up time point, results are given only in the secondary outcome section
Arm/Group | EM-10 Days Doxycycline | EM-doxycycline 15 Days | Controls
Number analyzed (Participants) | 108 | 117 | 81
number of participants
  number of patients with complete response | 79 | 85 | 81
  number of patients with NOIS | 7 | 6 | NA — Controls were not subjected to any intervention and were therefore not aplicable for evaluation on treatment outcome.

2. Secondary Outcome: Number of Patients (at 6 Months After Treatment With Doxycycline for 10 or 15 Days for Erythema Migrans) and Number of Control Subjects (Without a History of Lyme Borreliosis) With Nonspecific Symptoms.
Description: 6 months after treatment patients and controls were asked to complete a written questionnaire asking whether they had had any of 14 nonspecific symptoms (fatigue, malaise, arthralgias, headache, myalgias, pain in the spine, paresthesias, dizziness, nausea, insomnia, sleepiness, forgetfulness, concentration difficulties, or irritability) within the preceding week.
  For both patients and controls, the severity of each individual symptom was graded by the subject on a 10-cm visual analog scale (10 = most severe).
Time Frame: 6 months after treatment
Population: number of participants with nonspecific symptoms
Measure: Number; unit: number of participants
Groups:
- EM Patients: EM patients treated with doxycycline 100 mg b.i.d. for 10 or 15 days
- Controls: control subjects without a history of Lyme borreliosis
Arm/Group | EM Patients | Controls
Number analyzed (Participants) | 197 | 81
number of participants | 151 | 60

ADVERSE EVENTS:
Arm/Group | EM-10 Days Doxycycline | EM-doxycycline 15 Days | Controls
Serious Adverse Events (participants affected / at risk) | 24/108 | 32/117 | 0/0
Other Adverse Events (participants affected / at risk) | 5/108 | 9/117 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EM-10 Days Doxycycline (N=108) | EM-doxycycline 15 Days (N=117) | Controls (N=0)
Gastrointestinal symptoms, Photosensitivity (Gastrointestinal disorders) | 24 | 32 | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EM-10 Days Doxycycline (N=108) | EM-doxycycline 15 Days (N=117) | Controls (N=0)
Sleepiness, headache, vaginal discharge, dizziness, nervousness, obstipation (General disorders) | 5 | 9 | 0 (0)
sleepiness (General disorders) | 3 | 2 | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes